CLINICAL TRIAL: NCT06633094
Title: Home Management of Pediatric Buckle Fractures: Can Video Education Replace In-Person Visits?
Brief Title: Home Management of Pediatric Buckle Fractures
Acronym: HM-PBF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Peter J Apel, Orthopedic Hand and Upper Extremity Surgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1491
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Buckle Fracture; Patient Satisfaction
Keywords: Pediatric orthopedics; Distal radius fractures; Pediatric fractures; Fracture management; Patient education
MeSH Terms: conditions — Patient Satisfaction; Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person management (No Intervention): In-person group will be followed with standard-of-care clinic visits scheduled with an pediatric orthopaedic Surgeon at Carilion Clinic Institute for Orthopaedics and Neurosciences. Participants will complete a pediatric PROMIS assessment at baseline and 6 weeks for . Patients/guardians will complete a satisfaction survey.
- Home management (Experimental): Home-management group will be given access to an educational video explaining the nature of buckle fractures and treatment. all participants will enroll in MyChart to allow for asynchronous messages. Participants will complete a pediatric PROMIS assessment at baseline and 6 weeks. Patients/guardians will complete a satisfaction survey.
  Interventions: Other: Educational videos

INTERVENTIONS:
Other: Educational videos — Internet will be used to deliver educational videos to subjects enrolled in the home management arm of the study which will be available on the Carilion Clinic Orthopaedic Education YouTube Channel. This will consist of a prerecorded video made by the three pediatric orthopaedic surgeons on this study explaining the nature of buckle fractures and treatment. Participants will be sent a link to the video over email (an example of a similar video in clinical use at Carilion Orthopaedics and the script of the video can be found in the study document attached).
  Arms: Home management

SUMMARY:
The goal of this clinical trial is to determine if a home management plan incorporating video education can effectively replace in-person visits for children aged 7-17 diagnosed with distal radius buckle fractures.

The main questions it aims to answer are:

Is a home management plan with video education non-inferior to in-person management for patient satisfaction? Is a home management plan superior to in-person management for reducing healthcare-related time, missed work/school, inappropriate care (e.g., rigid casting), and healthcare resource consumption? Researchers will compare the home management group to the in-person management group to see if video education can reduce healthcare costs and the burden on patients without compromising care quality.

Participants will:

Be randomized to either the in-person group or the video-based home management group.

Complete a pediatric PROMIS assessment at baseline and 6 weeks. Complete a satisfaction survey at the conclusion of the study.

DETAILED DESCRIPTION:
Pediatric buckle fractures of the wrist are extremely common. In the U.S., these are often referred to a pediatric orthopaedic specialist, despite evidence that specialty follow-up is unnecessary. These unnecessary visits add to healthcare costs, especially for patients living in rural areas who must travel long distances to see specialists. Our group has been successful with short video-based education in prior work. In this study, the investigators aim to reduce the burden of care for buckle fracture patients and their parents/guardians. Our objective is to determine whether a home management plan centered around video education can replace in-person visits. Here, the investigators propose a prospective, randomized controlled non-inferiority study to determine if a home management plan incorporating video education can replace in-person visits for pediatric buckle fractures. This study has the potential to reduce the burden on patients and families who may have to travel long distances and miss school/work. In addition, this method of treatment has the potential to reduce healthcare costs and increase access for other patients with higher acuity medical needs.

Our current objective is to determine whether a home management plan centered around video education can effectively replace in-person visits.

Hypothesis 1: A home management plan for pediatric buckle fractures incorporating video education is non-inferior to in-person management for patient satisfaction.

Hypothesis 2: A home management plan for pediatric buckle fractures incorporating video education is superior to in-person management for time spent on healthcare activities, missed time from work, missed time from school, rate of inappropriate care (rigid casting and follow-up x-ray), level of health care resource consumption as measured by provider time spent on delivering care.

The investigators plan to perform a prospective, randomized controlled non-inferiority study to examine the effectiveness of educational videos on validated patient-reported outcomes.

Our study population will be composed of children who are diagnosed with a distal radius buckle fracture at Carilion Clinic. Subjects will be randomized to one of two groups: in-person management or home management through video education.

Incoming pediatric referrals containing the phrase: "distal radius fracture" "wrist fracture" or "buckle fracture" will be flagged and the x-rays will be reviewed within 4 business hours by one of the three pediatric orthopaedic surgeons on this study. If the fracture pattern meets inclusion criteria, the family will be offered the opportunity to enroll by the Clinical Research Coordinator/Clinical Research Assistant. Parent/guardians will acknowledge consent by secure electronic signature on REDCap. Children 7-17 years of age will be asked to assent.

Those randomized to the in-person group will meet with an Orthopaedic Surgeon at Carilion Clinic Institute for Orthopaedics and Neurosciences. the home management group will be given access to an educational video explaining the nature of buckle fractures and treatment. all participants will enroll in MyChart to allow for asynchronous messages. Participants from both groups will complete a pediatric PROMIS assessment at baseline and 6 weeks. Patients/guardians will complete a satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Any incoming pediatric orthopaedic referral containing the phrase: "distal radius fracture" "wrist fracture" or "buckle fracture
* A buckle fracture of the distal radius without opposite cortical break (an associated buckle fracture of the ulna is acceptable for inclusion)
* Age 5-17
* Access to a smartphone, tablet, or computer
* Access to internet to download or view videos

Exclusion Criteria:

* Other fractures
* Discontinuity of both cortices of the distal radius.
* Metabolic bone disease
* Developmental delay affecting assessment
* Inability to utilize technology to view videos or follow instructions
* Lack of internet or telephone access
* Family/caregiver inability to speak or read English or Spanish

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome Measurement Information System (PROMIS) Pediatric Short Form v2.0 - Physical Function Upper Extremity. | Baseline to 6 week follow-up
  This pediatric PROMIS assessment will be filled out at baseline and 6 weeks. All responses will be recorded within the study's REDCap database.
  Responses for each question:

SECONDARY OUTCOMES:
Parent Satisfaction Survey | Baseline to 6 week follow-up
  4 Questions:
  A survey will be sent to the parents/guardians to obtain the following information:
  1) Satisfaction with their care, measures on a 5-point Likert scale:
  * Participants will select: Strongly Disagree, Disagree, Neither Agree or Disagree, Agree, or Strongly Agree 2) Time spent on healthcare activities
  * Recorded in minutes 3) Time missed from work
  * Recorded in minutes 4) Time missed time from school.
  * Recorded in minutes
Rigid Casting | Baseline to 6 week follow-up
  Electronic medical record chart review will be performed to determine:
  Rate of rigid casting
  - Yes or No
Rate of follow-up X-rays | Baseline to 6 week follow-up
  Electronic medical record chart review will be performed to determine: Number of x-rays ordered during follow-up care
Provider time spent on delivering care | Baseline to 6 week follow-up
  Electronic medical record chart review will be performed to determine: Number of follow-up visits (minutes per session)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Apel, MD, PhD, Principal Investigator — Carilion Clinic Orthopaedic Surgery
Locations (1):
- Carilion Clinic Orthopaedic Surgery, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landin LA. Epidemiology of children's fractures. J Pediatr Orthop B. 1997 Apr;6(2):79-83. doi: 10.1097/01202412-199704000-00002. PMID 9165435
- [Background] Bae DS, Howard AW. Distal radius fractures: what is the evidence? J Pediatr Orthop. 2012 Sep;32 Suppl 2:S128-30. doi: 10.1097/BPO.0b013e31824b2545. PMID 22890451
- [Background] Baig MN, Egan C. Improving Management of Paediatric Buckle Fracture in Orthopaedic Outpatients: A Completed Audit Loop. Cureus. 2017 Nov 8;9(11):e1829. doi: 10.7759/cureus.1829. PMID 29326858
- [Background] Koelink E, Boutis K. Paediatrician office follow-up of common minor fractures. Paediatr Child Health. 2014 Oct;19(8):407-12. doi: 10.1093/pch/19.8.407. PMID 25382996
- [Background] Symons S, Rowsell M, Bhowal B, Dias JJ. Hospital versus home management of children with buckle fractures of the distal radius. A prospective, randomised trial. J Bone Joint Surg Br. 2001 May;83(4):556-60. doi: 10.1302/0301-620x.83b4.11211. PMID 11380131
- [Background] Firmin F, Crouch R. Splinting versus casting of "torus" fractures to the distal radius in the paediatric patient presenting at the emergency department (ED): a literature review. Int Emerg Nurs. 2009 Jul;17(3):173-8. doi: 10.1016/j.ienj.2009.03.006. Epub 2009 May 7. PMID 19577205
- [Background] Boutis K. Common pediatric fractures treated with minimal intervention. Pediatr Emerg Care. 2010 Feb;26(2):152-7; quiz 158-62. doi: 10.1097/PEC.0b013e3181ce310c. PMID 20145510
- [Background] Koelink E, Schuh S, Howard A, Stimec J, Barra L, Boutis K. Primary Care Physician Follow-up of Distal Radius Buckle Fractures. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-2262. Epub 2015 Dec 10. PMID 26729537
- [Background] Plint AC, Perry JJ, Correll R, Gaboury I, Lawton L. A randomized, controlled trial of removable splinting versus casting for wrist buckle fractures in children. Pediatrics. 2006 Mar;117(3):691-7. doi: 10.1542/peds.2005-0801. PMID 16510648
- [Background] Davidson JS, Brown DJ, Barnes SN, Bruce CE. Simple treatment for torus fractures of the distal radius. J Bone Joint Surg Br. 2001 Nov;83(8):1173-5. doi: 10.1302/0301-620x.83b8.11451. PMID 11764434
- [Background] Williams BA, Palumbo NE, Phillips SA, Blakemore LC. What They Want - Caregiver and Patient Immobilization Preferences for Pediatric Buckle Fractures of the Wrist. Iowa Orthop J. 2020;40(1):83-90. PMID 32742213
- [Background] Heikkinen K, Helena LK, Taina N, Anne K, Sanna S. A comparison of two educational interventions for the cognitive empowerment of ambulatory orthopaedic surgery patients. Patient Educ Couns. 2008 Nov;73(2):272-9. doi: 10.1016/j.pec.2008.06.015. PMID 18678461
- [Background] Wright JE, Brown RR, Chadwick C, Karadaglis D. The use of the Internet by orthopaedic outpatients. J Bone Joint Surg Br. 2001 Nov;83(8):1096-7. doi: 10.1302/0301-620x.83b8.12390. No abstract available. PMID 11764418
- [Background] Yi PH, Ganta A, Hussein KI, Frank RM, Jawa A. Readability of arthroscopy-related patient education materials from the American Academy of Orthopaedic Surgeons and Arthroscopy Association of North America Web sites. Arthroscopy. 2013 Jun;29(6):1108-12. doi: 10.1016/j.arthro.2013.03.003. PMID 23726111
- [Background] Cotugna N, Vickery CE, Carpenter-Haefele KM. Evaluation of literacy level of patient education pages in health-related journals. J Community Health. 2005 Jun;30(3):213-9. doi: 10.1007/s10900-004-1959-x. PMID 15847246
- [Background] Bini SA, Schilling PL, Patel SP, Kalore NV, Ast MP, Maratt JD, Schuett DJ, Lawrie CM, Chung CC, Steele GD. Digital Orthopaedics: A Glimpse Into the Future in the Midst of a Pandemic. J Arthroplasty. 2020 Jul;35(7S):S68-S73. doi: 10.1016/j.arth.2020.04.048. Epub 2020 Apr 22. PMID 32416956
- [Background] Colaco K, Willan A, Stimec J, Barra L, Davis A, Howard A, Boutis K. Home Management Versus Primary Care Physician Follow-up of Patients With Distal Radius Buckle Fractures: A Randomized Controlled Trial. Ann Emerg Med. 2021 Feb;77(2):163-173. doi: 10.1016/j.annemergmed.2020.07.039. Epub 2020 Oct 21. PMID 33500115